CLINICAL TRIAL: NCT06082336
Title: Prospective Clinical Performance Evaluation of the In-Vitro Diagnostics Medical Device MaGIA IBC for the CombIned screENing of HIV, Hepatitis B and Hepatitis C
Acronym: MAGICIEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MagIA Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MAGIA-IBC-EP-01
Record Dates: First submitted 2023-10-02; First posted 2023-10-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Combined Point of Care Diagnostic of HIV, HBV and HCV
Keywords: point of care diagnostic; HIV; HCV; HBV
MeSH Terms: conditions — Hepatitis B; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): This study is single arm.
  Interventions: Diagnostic Test: MagIA IBC test in capillary blood; Diagnostic Test: MagIA IBC test in other blood matrices

INTERVENTIONS:
Diagnostic Test: MagIA IBC test in capillary blood — After a finger prick, patients will be taken a drop of capillary drop. This drop will be used to perform the MagIA IBC test.
Diagnostic Test: MagIA IBC test in other blood matrices — Blood samples will be taken and used to perform the MagIA IBC in veinous blood, serum and plasma, except for outdoor tested subjects

SUMMARY:
Prospective, cross-sectional, adaptative study to evaluate the clinical performance of the In-Vitro Diagnostics Medical Device MagIA IBC (a Multiplex Point-of-Care Test for the detection of HIV, HBV and HCV) in detecting anti-HIV antibodies (HIV-Ab), anti-HCV antibodies (HCV-Ab), and HBs antigens (HBs-Ag) in serum, plasma, venous blood and capillary blood. If not prescribed for the patient care, blood drawings, and finger pricks will be performed on the patient for the purpose of the clinical study.

The Study includes a Technical Adjustment Phase (to identify optimized acquisition parameters and to define the decision threshold for the diagnostic) followed by a Validation Phase (to validate the concordance between the matrices and to evaluate the Specificity and the Sensibility of the diagnostics).

Validation Phase is between Sept. 2024 and still ongoing.

ELIGIBILITY:
Inclusion Criteria:

IC1. A Male or Female aged of at least 18 years

IC2. A person responding to one of the following conditions:

* known having HIV infection
* or known having HBV infection
* or known or suspected having HCV infection with anti-HCV RDT positive. IC3. A person having given consent to participate the study, IC4. A person covered by a medical insurance or being enrolled during an outdoor testing campaign.

Exclusion Criteria:

EC1. A person for whom blood sampling would represent a risk, EC2. A person protected by law (minor, under guardianship or curatorship, childbearing, or breastfeeding female, hospitalized without consent, under administrative or judicial supervision)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Clinical Performance of the MagIA IBC test in determining the serological status of HIV infection, HCV infection (current infection only) and HBV infection | baseline
  For each of the 3 diagnostics, the corresponding Endpoints are the Sensitivity (Se) and Specificity (Sp) of MagIA IBC.

SECONDARY OUTCOMES:
Concordance of the results delivered by MagIA IBC for HIV and HBV, on each of the selected matrices (i.e. serum, plasma, venous and capillary blood). | baseline
  For HIV and HBV, the corresponding Endpoint is the Kappa coefficient calculated for each of the 6 concordance tables comparing the results in the selected matrices.
Adverse events of MagIA IBC test | 1 day
  Adverse events will be collected to assess safety of the device.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Européen de Marseille, Marseille, France
  - Centre Hospitalier de Perpignan - Equipe Mobile Hépatites, Perpignan

IPD SHARING:
Plan to Share IPD: Undecided